CLINICAL TRIAL: NCT04430686
Title: Respiratory Complications Associated With ALS and Their Treatments
Brief Title: Respiratory Complications in ALS
Status: Completed | Type: Observational
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: REC:20/L0/0275
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Motor Neuron Disease; Pneumonia
MeSH Terms: conditions — Motor Neuron Disease; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionaires — Any validated functional rating scale, such as the Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS) or the ALSFRS-Revised (if available)

SUMMARY:
Respiratory failure is the leading cause of death in motor neuron disease (MND) patients. Symptoms of respiratory dysfunction in MND patients include sleep disturbance, excessive daytime somnolence, morning headaches and cognitive changes. Almost all MND patients will develop respiratory problems during the course of their disease. In a small percentage of MND patients, respiratory failure may present as the primary symptom at onset, whereas more commonly it develops later in the disease.

DETAILED DESCRIPTION:
Respiratory failure is the leading cause of death in motor neuron disease (MND) patients. Symptoms of respiratory dysfunction in MND patients include sleep disturbance, excessive daytime somnolence, morning headaches and cognitive changes. Almost all MND patients will develop respiratory problems during the course of their disease. In a small percentage of MND patients, respiratory failure may present as the primary symptom at onset, whereas more commonly it develops later in the disease. (1) Forced vital capacity (FVC), taken either supine or erect, is the most commonly used measurement tool of respiratory function. Such measures are well recognized predictors of survival (2), with supine FVC a more accurate marker of diaphragmatic weakness (1). However, FVC may not be sensitive for the detection of early respiratory failure and can be technically difficult to perform in patients with severe bulbar weakness (3). Other respiratory measures include maximal inspiratory pressure (MIP), maximal expiratory pressure (MEP), sniff nasal inspiratory pressure (SNIP) and, less commonly, formal assessment of arterial blood gases (ABG). Interpretation of the trends of these measures over time, combined with the clinical picture, determines appropriate respiratory management. Significantly, the advent of non-invasive ventilation (NIV) has provided clear benefit in terms of improving symptoms, QOL and prolonging survival by up to 7 months in MND patients, making NIV a central armamentarium of respiratory management in these patients (4) Bilevel ventilation devices (Bi-PAP) are most commonly used as initial therapy. There are no established evidence-based guidelines regarding optimal timing for initiation of NIV.Some studies suggest that an early introduction of NIV may increase survival (5), reduce respiratory-related energy expenditure (6) and improve adherence to therapy and QOL (7).Once initiated, poor optimisation of NIV represents an independent risk factor for mortality (8) However, there are no randomized control trial data available that have compared the specific parameters of bilevel modes of ventilation across various patient cohorts. Different strategies have been used to optimize patient comfort, including adjusting the type of mask and fittings, providing humidified air and testing different Bi-PAP pressure settings. Despite these measures, up to 30% of MND patients cannot tolerate therapy due to secondary effects of anxiety, emotional lability from pseudobulbar palsy, excessive salivation, claustrophobia and nasal bridge soreness (8) Importantly, the key factors that affect overall compliance with this treatment are the presence of bulbar dysfunction with bulbar onset patients six times less likely to tolerate NIV than those with limb onset disease (9) Future efforts must be focused on determining more accurate testing for early respiratory failure, optimal time to initiate NIV and the comfortable adaptation of NIV devices for patients with bulbar weakness

ELIGIBILITY:
Inclusion Criteria:

Patients with ALS

Exclusion Criteria:

None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population with ALS
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Overall survival after initiation of assisted ventilation | 1 year

SECONDARY OUTCOMES:
Survival at one month and six months or longer | 1 month and 6 months
Quality of life assessed using validated health status questionnaires | 1 year
  Any validated functional rating scale, such as the Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS) or the ALSFRS-Revised (if available)
Time of initiation of diagnosis of MND and initiation of NIV | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- LiverpoolUHNHS, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We will make the research available to any MND researchers/patients